CLINICAL TRIAL: NCT00094068
Title: A Pilot Study to Detect the Effect of Sildenafil Citrate on Cerebral Blood Perfusion in Multiple Sclerosis Patients by Perfusion MRI
Brief Title: The Effect of Sildenafil Citrate (Viagra® (Registered Trademark)) on Brain Blood Flow in Multiple Sclerosis Patients
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050003; 05-CC-0003
Record Dates: First submitted 2004-10-09; First posted 2004-10-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Multiple Sclerosis
Keywords: Gray Matter; White Matter; Cerebral Blood Flow; Cerebral Blood Volume; Lesion; MRI; Multiple Sclerosis; Perfusion; Imaging; Sildenafil; MS; Healthy Volunteer; HV
MeSH Terms: conditions — Multiple Sclerosis

SUMMARY:
This study will determine whether sildenafil citrate, commonly known as Viagra, can cause increased blood flow to the brain in a wide range of multiple sclerosis (MS) patients, including women. Although people with MS can have reduced blood flow in the brain as part of the disease process, it has been observed that men with MS may have increased blood flow to the brain while taking sildenafil citrate. This study will measure brain blood flow or blood volume in men and women with MS before and after taking Viagra and compare the results to those in healthy volunteers in an effort to better understand the disease.

Healthy volunteers 18 years of age and older and patients with MS between 18 and 55 years of age may be eligible for this study. Volunteers are screened with a medical history and physical examination, and patients with MS are evaluated with a complete neurological examination and screening for heart disease, including history of chest pain, heart attack, and use of nitrates.

Participants undergo magnetic resonance imaging (MRI) before and after taking Viagra. During the scanning, subjects lie still on a table that can slide in and out of the cylindrical metal scanner. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. First, a scan is obtained of the carotid arteries (major arteries in the neck supplying blood to the brain) to determine if the arteries are narrowed, and then baseline MRI scans and measures of brain blood flow are obtained. The subject then comes out of the scanner and takes a Viagra pill. After 1 hour, the subject returns to the scanner and more scans are obtained to determine changes in brain blood flow and blood volume following Viagra.

A catheter (thin plastic tube) is placed in the subject's arm before he or she enters the magnet for the second time for injection of a contrast agent called gadolinium DTPA, which allows brain structures to be distinguished more clearly.

DETAILED DESCRIPTION:
Advances in MR perfusion imaging have provided clinical researchers with the opportunity to quantify regional cerebral blood flow (CBF). It has been shown that cerebral perfusion in patients with multiple sclerosis (MS) is reduced, particularly in the grey matter. However, preliminary data in a small number of male secondary progressive (SP) MS patients with erectile dysfunction suggests that sildenafil citrate (Viagra® (Registered Trademark)) helps to increase grey matter perfusion. The purpose of this study is to extend these findings to male MS patients without erectile dysfunction and female MS patients by comparing CBF measures of MS patients of both sexes, to age and gender-matched healthy controls. CBF will be measured before and one hour after taking sildenafil citrate.

ELIGIBILITY:
INCLUSION CRITERIA:

Any healthy normal volunteer above the age of 18 who is capable of giving informed consent recruited or self referred through the NIH Volunteer office will be eligible for this study.

All healthy normal volunteers will be included as long as there is no recorded or documented signs or symptoms of CNS disease, contraindications to a MRI and have a "normal age appropriate" MRI of the brain.

Patients seen in the Neuroimmunology MS clinic with a confirmed diagnosis of Multiple Sclerosis based upon previous history of two clinical neurological attacks separated in time and in spatial location or combination of Clinical and MRI findings of a single enhancing lesion in the brain or spine along with multiple T2 hyperintensities in the juxtacortical, periventricular or infratentorial white matter according to the McDonald criteria will be included in this study.

Relapsing-remitting or secondary progressive MS who have had more than one relapse within 18 months preceding study enrollment will be recruited from the MS 7th floor clinic in the NINDS at the NIH. MS patients will have EDSS score between 1.0 - 6.5, inclusive. MS patients seen and treated in the NINDS MS clinic are representative of the general MS population that is Female: male ratio of approximately 3:2, Caucasian and African American, between ages of 18-55 years old.

Give written informed consent prior to any testing under this protocol, including screening/pre-treatment tests and evaluations that are not considered part of the patient's routine care.

EXCLUSION CRITERIA:

Healthy Controls and MS patients will be excluded if they have contraindications to MR scanning, such as the following:

1. aneurysm clip
2. implanted neural stimulator
3. implanted cardiac pacemaker or autodefibrillator
4. cochlear implant
5. ocular foreign body (e.g., metal shavings)
6. insulin pump

Healthy controls and MS patients will be excluded from this study if they have the following:

1. History of heart attack
2. History of treatment with nitrates for heart condition
3. History of carotid artery stenosis or evidence of greater than 50% carotid stenosis on screening MR angiogram
4. History of known vascular disease
5. History of stroke
6. History of migraine
7. Subjects who have a history of a reaction to MR contrast agents specifically gadopentetate dimeglumine will be excluded from participating in the contrast agent administration part of this protocol.
8. Healthy controls will be excluded if have history of alcohol or drug abuse.
9. Healthy controls will be excluded if Concurrent, clinically significant (as determined by the investigator) gastrointestinal, immunologic, pulmonary, neurologic, renal, and/or other major disease.
10. Healthy controls will be excluded if they have a previous known abnormality on Brain MRI examination.
11. Pregnant and lactating women will be excluded from the study.
12. Since certain drugs may interfere with the ability of the vessels in your brain to respond to Viagra, subjects taking steroids or sildenafil (within 24 hours) will be excluded from this study.

MS patients will also be excluded from study entry if any of the following exclusion criteria exist at the time of enrollment:

1. Pregnant and lactating women who are MS patients will be excluded from the study.
2. Diagnosis of primary progressive MS, defined as gradual progression of disability from the onset without relapses.
3. Concurrent, clinically significant (as determined by the investigator) immunologic, pulmonary, gastrointestinal, neurologic, renal, and/or other major disease in MS patients.

Treatment History in MS patients

If prior treatment with steroids was received, the subject must have been off treatment for the required period prior to enrollment (see below).

Agent: Corticosteroids

Time Required off Agent Prior to Enrollment: 8 weeks

Unwillingness or inability to comply with the requirements of this protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's returning for follow-up visits to the NINDS, Neuroimmunology Clinic will be sufficient reason to exclude a subject.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76
Dates: Start 2004-10; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Lublin FD, Reingold SC. Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology. 1996 Apr;46(4):907-11. doi: 10.1212/wnl.46.4.907. PMID 8780061
- [Background] Prineas J. Pathology of the early lesion in multiple sclerosis. Hum Pathol. 1975 Sep;6(5):531-54. doi: 10.1016/s0046-8177(75)80040-2. PMID 170186
- [Background] van der Valk P, De Groot CJ. Staging of multiple sclerosis (MS) lesions: pathology of the time frame of MS. Neuropathol Appl Neurobiol. 2000 Feb;26(1):2-10. doi: 10.1046/j.1365-2990.2000.00217.x. PMID 10736062